CLINICAL TRIAL: NCT00223522
Title: Do Self-Report and Physician Impressions of Adherence to Oral Antipsychotic Medication Agree With Objective Data?
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Other Study IDs: 034-0013-002; 034-0013-002
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Schizoaffective
Keywords: Schizophrenia; Schizoaffective; MEMS; adherence to antipsychotic medication
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: MEMS caps

SUMMARY:
The purpose of this study is to prospectively examine adherence to oral atypical antipsychotics in patients with schizophrenia. We are psrticularly interested in examining the level of agreement among self-report, physician impressions and objective measures of adherence. We believe that physicians, casemanagers, and clients significantly overestimate the level of adherence.

DETAILED DESCRIPTION:
Fifty schizophrenia patients will be recruited at the time of their clinic visit to Tri-County MHMR Services and the El Paso Community MHMR Center. Both physicians and patients will be asked to rate the patient's medication adherence on their index clinic visit. Initial ratings will also occur at this visit. After filling their medication prescription, all subjects will be given electronic medication caps that record each time and date their medication container is opened. Patients will then be followed in the community for the next 12 weeks to observe actual adherence to medication from the index visit to the next successive clinic visit. Every two weeks pills will be counted and data will be retrieved from the electronic medication caps. During the first and last two weeks of study, blood will be sampled on two randomly selected occasions approximately 72 hours apart. Self-report and physician assessment of adherence, symptom and attitudinal measures will be obtained a second time at the second clinic visit 12 weeks after the index visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia or Schizoaffective disorder
* Between the ages of 18-55
* no documented history of head injury, mental retardation or neurological disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2004-04; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I Velligan, Ph.D., Principal Investigator — University of Texas
Locations (1):
- UTHSCSA, San Antonio, Texas, United States